CLINICAL TRIAL: NCT02986984
Title: Transformative Research In DiabEtic NephropaThy
Acronym: TRIDENT
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: MOUNT SINAI HOSPITAL (Other); University of North Carolina (Other); Northwestern University (Other); University of New Mexico (Other); Stanford University (Other); The University of Texas Health Science Center at San Antonio (Other); Ohio State University (Other); Yale University (Other); Albert Einstein College of Medicine (Other); Oregon Health and Science University (Other); Lehigh Valley Health Network (Other); University of Arkansas (Other); University of Southern California (Other); University of Virginia (Other); Regeneron Pharmaceuticals (Industry); Boehringer Ingelheim (Industry); GlaxoSmithKline (Industry); Gilead Sciences (Industry); Juvenile Diabetes Research Foundation (Other); Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: 824503
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Diabetic Nephropathies; Diabetic Glomerulosclerosis
Keywords: Diabetes; Chronic kidney disease; Progression; Genomics; Transcriptomics
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus; Renal Insufficiency, Chronic; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buffy Coat (Germline DNA) Kidney Biopsy Cores Urine and blood aliquots for RNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Confirmed Diabetic Nephropathy: Patients undergoing a clinically indicated kidney biopsy with a history of diabetes who satisfy pre-specified criteria for diabetic nephropathy.
  Interventions: Other: There is no intervention
- Confirmed Non-diabetic Nephropathy: Patients undergoing a clinically indicated kidney biopsy with a history of diabetes who fail pre-specified criteria for diabetic nephropathy.
  Interventions: Other: There is no intervention

INTERVENTIONS:
Other: There is no intervention — There are no interventions
  Other Names: There are no interventions

SUMMARY:
This is a prospective, observational, cohort study of patients with a clinical diagnosis of diabetes who are undergoing clinically indicated kidney biopsy. The intent is to collect, process, and study kidney tissue and to harvest blood, urine and genetic materials to elucidate molecular pathways and link them to biomarkers that characterize those patients have a rapid decline in kidney function (> 5 mL/min/1.73m2/year) from those with lesser degrees of kidney function change over the period of observation. High through-put genomic analysis associated with genetic and biomarker testing will serve to identify key potential therapeutic targets for DKD by comparing patients with rapid and slow progression patterns. Each participating clinical site will search for, consent, harvest the biopsy sample, and enroll the participants as required for the TRIDENT protocol.

DETAILED DESCRIPTION:
Progress in the area of diabetic kidney research leading to new therapeutics development has been very limited. Indeed, no new medicines indicated for the treatment of chronic kidney disease (CKD) have been approved since ARB's have become standard of care nearly 15 years ago. Several factors explain the limited progress including but not limited to; a) animal and cell culture models do not recapitulate human DKD b) human genetic studies so far have failed to identify reproducible genetic variants associated with DKD c) the clinical manifestation of DKD is heterogeneous and might have even changed since the original description d) DKD is a clinical diagnosis and it is not clear what percentage of patients have histological disease.

Laboratory mice have served as invaluable tools to understand human disease development. As mouse genetic tools became readily available, it enabled us to perform time and cell type specific gene manipulation in animals to generate disease models and to understand the contributions of specific pathways. Unfortunately, mouse models do not recapitulate human diabetic kidney disease as animals develop only early DKD lesions; mesangial expansion and mild albuminuria11. Most models do not develop arterial hyalinosis, tubulointerstitial fibrosis and declining glomerular filtration rate (GFR); hallmarks of progressive DKD. There are several fundamental differences in gene expression patterns and physiology of human and murine kidneys. Such differences may explain the lack of translatability between mice and humans of pharmacological approaches aimed at treating DKD. This seems to be a general trend in other disease areas as well (for example Alzheimer's disease), leading to a recent movement toward translational and clinical research with increasing reliance on human samples.

Human genetic studies made paradigm-shifting observations in relatively rare monogenic forms of kidney diseases (including polycystic kidney disease and focal segmental glomerulosclerosis). Diabetic CKD on the other hand follows a complex polygenic pattern. Currently, the most powerful method to define the genetics of complex diseases such as DKD is genome wide association (GWAS), where associations between polymorphisms and the disease state are tested. Prior studies indicate that for complex traits, such as DKD, genetic polymorphisms that are associated with disease state are localized to the non-coding region of the genome12,13. Moreover, the genetic architecture of diabetic kidney disease has not been characterized and several large collaborations are currently addressing this issue14. Thus, the next challenge is to define target genes, target cell types and the mode of dysregulation caused by non-coding snips (SNPs15). Such studies require large collection of human tissue samples from disease relevant organs.

Diabetic kidney disease (DKD) remains a clinical diagnosis. Subjects with CKD in the presence of diabetes and albuminuria are considered to have diabetic nephropathy. Such definition is used in clinical practice and in research studies including clinical trials. Studies performed in 1980 provide the basis for the practice16,17. Investigators stage DKD as a progressive disease, beginning with the loss of small amounts of albumin into the urine (30-300mg/day; known as the stage of microalbuminuria, high albuminuria, occult or incipient nephropathy), then larger amounts (>300mg/day; known as macroalbuminuria, very high albuminuria or overt nephropathy), followed by progressive decline in kidney function (eGFR), renal impairment and ultimately ESRD 17-19. This paradigm has proved useful in clinical studies, especially in type 1 diabetes, for identifying cohorts at increased risk of adverse health outcomes. However, boundaries between stages of DKD are artificial and the relationship between urinary albumin excretion and adverse health outcomes is log-linear in clinical practice. Indeed, the American Diabetes Association recently abandoned staging of albuminuria (ACR) for a more-straightforward [ACR >30 mg/g, (albuminuria present); ACR <30 mg/g (albuminuria absent)] criterion. Moreover, many patients, and especially those with type 2 diabetes, do not follow this classical course in modern clinical practice. For example, many subjects with DKD do not manifest excessive urinary albumin loss20. Indeed, of the 28% of the UKPDS cohort who developed moderate to severe renal impairment, half did not have preceding albuminuria. In the Diabetes Control and Complications Trial (DCCT), of the 11% patients with type 1 diabetes who developed an eGFR<60 ml/min/1.73m2, 40% never had experienced overt nephropathy21. In addition, most patients with microalbuminuria do not progressively exhibit an increase in urinary albumin excretion as in the classical paradigm with treatment-induced and spontaneous 'remission' of albuminuria widely observed22,23. Consequently, individuals with microalbuminuria may better be regarded as being at increased risk of developing progressive renal disease (as well as cardiovascular disease and other diabetic complications), rather than as actually having DKD per se. While over the last 40 years it became evident that the original description of DKD needs revision, no alternative criteria have emerged given the lack of solid data on the correlation between histopathological (gold standard) DKD diagnosis and clinical manifestations. It is also possible that, with the introduction of better glycemic control and anti-renin (RAAS) blockade, the disease has evolved necessitating new observational cohorts to understand the clinical disease course and manifestations.

Diabetic kidney disease presents with a variable rate of kidney function decline24. Data from large observational cohorts indicate that GFR decline frequently does not follow a linear course. Several groups are working on modeling GFR decline patterns in patients. Such studies contributed to emphasizing patients termed as "rapid progressors". There is no consensus definition for rapid progression. Many studies define rapid progressors as patients with greater than 3 cc/year GFR decrease but alternative cut points such as even 10 cc/year has also been used. Identification and clinical characterization of rapid progressors became the center of several large scale efforts as these are the patients who would likely need intensive clinical management25. Furthermore recent post-hoc analyses of the Diabetic Nephropathy (IDNT and RENAAL) studies indicate that clinical trial outcomes are mostly driven by a small number of subjects with unusually rapidly progressive GFR decline i.e. subjects that display characteristics of rapid progressors. While investigators are still awaiting accurate descriptions, biomarker and clinical descriptive studies have yielded several interesting observations. Albuminuria remains one of the strongest risk factor for "FDA-approved" (hard) renal outcomes; doubling of serum creatinine, dialysis or death. Indeed some of the latest studies indicate that using a 4 or a 6 variable model, that includes albuminuria, age, sex, serum phosphate, serum calcium and serum albumin has C-statistics score of 0.84-0.91 to predict ESRD 26,27. During the last years several new biomarkers have been identified that can potentially identify patients who are at increased risk for rapid loss of kidney function. For example blood and urinary levels of kidney injury molecule (KIM1) shows promise to identify patients who are at risk for kidney function decline. Recently, investigators showed that circulating levels of tumor necrosis factor receptor 1 and 2 levels can identify patients with rapidly declining renal function 28. While these markers are generating increased interest; the critical questions remains; why do some patients follow a rapid decline in kidney function?

ELIGIBILITY:
Inclusion Criteria:

* Type 1 and 2 Diabetes by American Diabetes Association (ADA) criteria
* Willingness to comply with study requirements, including intention to fully participate in protocol-specified follow-up at a clinical study site
* Able to provide informed consent
* Adult participants
* Planned medically indicated kidney biopsy, prescribed by a practicing nephrologist

Exclusion Criteria:

* End Stage Renal Disease (ESRD), defined as chronic dialysis or kidney transplant
* History of receiving dialysis for more than 30 days prior to biopsy
* Institutionalized
* Solid organ or bone marrow transplant recipient at time of first kidney biopsy
* Less than 3-year life expectancy
* History of active alcohol and/or substance abuse that in the investigator's assessment would impair the subject's ability to comply with the protocol
* Unable to provide informed consent
* Evidence of active cancer requiring treatment, other than non-melanoma skin cancer

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (18 years of age and older) with diabetes who are scheduled to have a clinically-indicated kidney biopsy.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Rapid progression of kidney function loss | up to three years
  • Identification of epigenetic, genetic, renal, genomic, and biomarker profiles that differentiates patients with rapid GFR decline (>5cc/min) from those with slower (<5cc/min) rate of progression.

SECONDARY OUTCOMES:
Serious Adverse Events | up to three years
  Prolonged hospitalization or need for intervention after kidney biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Katalin Susztak, MD, Principal Investigator — University of Pennsylvania
Locations (17):
- United States (17):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of Southern California, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - Northwestern University, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - Mount Sinai Hospital, New York, New York
  - Columbia University, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Townsend RR, Guarnieri P, Argyropoulos C, Blady S, Boustany-Kari CM, Devalaraja-Narashimha K, Morton L, Mottl AK, Patel U, Palmer M, Ross MJ, Sarov-Blat L, Steinbugler K, Susztak K; TRIDENT Study Investigators. Rationale and design of the Transformative Research in Diabetic Nephropathy (TRIDENT) Study. Kidney Int. 2020 Jan;97(1):10-13. doi: 10.1016/j.kint.2019.09.020. No abstract available. PMID 31901339
- [Result] Abedini A, Zhu YO, Chatterjee S, Halasz G, Devalaraja-Narashimha K, Shrestha R, S Balzer M, Park J, Zhou T, Ma Z, Sullivan KM, Hu H, Sheng X, Liu H, Wei Y, Boustany-Kari CM, Patel U, Almaani S, Palmer M, Townsend R, Blady S, Hogan J, Morton L, Susztak K; TRIDENT Study Investigators. Urinary Single-Cell Profiling Captures the Cellular Diversity of the Kidney. J Am Soc Nephrol. 2021 Mar;32(3):614-627. doi: 10.1681/ASN.2020050757. Epub 2021 Feb 2. PMID 33531352
- [Result] Palmer MB, Abedini A, Jackson C, Blady S, Chatterjee S, Sullivan KM, Townsend RR, Brodbeck J, Almaani S, Srivastava A, Avasare R, Ross MJ, Mottl AK, Argyropoulos C, Hogan J, Susztak K. The Role of Glomerular Epithelial Injury in Kidney Function Decline in Patients With Diabetic Kidney Disease in the TRIDENT Cohort. Kidney Int Rep. 2021 Feb 3;6(4):1066-1080. doi: 10.1016/j.ekir.2021.01.025. eCollection 2021 Apr. PMID 33912757
- [Result] Hogan JJ, Owen JG, Blady SJ, Almaani S, Avasare RS, Bansal S, Lenz O, Luciano RL, Parikh SV, Ross MJ, Sharma D, Szerlip H, Wadhwani S, Townsend RR, Palmer MB, Susztak K, Mottl AK; TRIDENT Study Investigators. The Feasibility and Safety of Obtaining Research Kidney Biopsy Cores in Patients with Diabetes: An Interim Analysis of the TRIDENT Study. Clin J Am Soc Nephrol. 2020 Jul 1;15(7):1024-1026. doi: 10.2215/CJN.13061019. Epub 2020 Apr 27. No abstract available. PMID 32341009